CLINICAL TRIAL: NCT01159821
Title: An Open-Label Study to Assess the Effect of CYP2D6 Inhibitor Paroxetine on the Single-Dose Pharmacokinetics of JNJ-31001074 in Healthy Subjects
Brief Title: A Drug Interaction Study of 31001074 and Paroxetine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CR017242; 31001074ATT1014 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: 31001074; Paroxetine; CYP2D6 inhibitor
MeSH Terms: interventions — Paroxetine

ARMS (1):
- 001 (Experimental): 31001074/paroxetine 1 tablet of 31001074 will be administered on Day 1 and Day 13. One 20-mg paroxetine tablet will be administered once daily from Days 4 through 15
  Interventions: Drug: 31001074/paroxetine

INTERVENTIONS:
Drug: 31001074/paroxetine — 1 tablet of 31001074 will be administered on Day 1 and Day 13. One 20-mg paroxetine tablet will be administered once daily from Days 4 through 15

SUMMARY:
The purpose of this study is to determine the concentration of 31001074 in blood samples from healthy volunteers who have been administered 31001074 and paroxetine.

DETAILED DESCRIPTION:
This is an open-label (both volunteer and study physician will know the identity of study treatment) pharmacokinetic study to determine the effects, if any that multiple 20-mg doses of paroxetine have on the concentration of a single dose of study drug (referred to as 31001074) in the bloodstream after paroxetine and 31001074 are administered orally (by mouth) to healthy adult volunteers. Paroxetine is an approved drug used to treat patients with psychiatric disorders and 31001074 is a drug that is currently under development for potential uses in the treatment of patients with nervous system disorders. Approximately 14 healthy volunteers will participate in the study for approximately 45 days (includes a screening period of up to 29 days to determine eligibility and a 16 day treatment period). Volunteers will be required to stay overnight at the study center during the 16-day treatment period. During the 16-day treatment period, volunteers will receive 2 doses of 31001074 and 12 doses of paroxetine. At Screening, a blood sample will be collected from all volunteers for pharmacogenomic analysis (ie, genetic testing) to identify volunteers genetically-determined to have high activity of an enzyme (CYP2D6) that is involved in the processing of 31001074 by the body. Additional blood samples will be obtained from volunteers at protocol-specified time points during the study to determine the concentration of 31001074 and paroxetine in plasma (the colorless portion of blood). Safety will be evaluated during the study by monitoring adverse events (side effects) reported and findings from clinical laboratory tests, vital signs measurements, electrocardiograms (ECGs), and physical examinations performed. In addition, volunteers will be instructed to report the occurrence of adverse events that are considered by the study physician to be serious (as defined by the protocol) for up to 30 days after the administration of the last dose of study drug. A single dose of 31001074 will be administered on Day 1 and Day 13 (total 2 doses). Paroxetine will be administered once daily from Days 4 through 15 (total 12 doses). All doses, including 31001074 and paroxetine will be administered at the same time (approximately 8 am), except on Day 13, when paroxetine will be administered 30 minutes (approximately 7:30 am) before the administration of 31001074.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) (weight [kg]/height2 [m]2) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Have a blood pressure after the healthy volunteer is supine [ie, lying down face up] for 5 minutes between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic at screening and at admission to the study center on Day -1
* If a woman, must be of nonchildbearing potential, i.e., postmenopausal (no spontaneous menses for at least 2 years) or surgically sterile
* Be a nonsmoker

Exclusion Criteria:

* Have a history of or a current medical illness that the investigator (study physician) considers to be clinically significant, a history of chronic uveitis (inflammation of the eye persisting for a long time) or any any intraocular surgery (except for cataract extraction, laser in situ keratomileusis [LASIK], or photorefractive keratectomy [PRK] procedures [ie, procedures used to reshape the cornea of the eye])
* Have clinically significant abnormal laboratory values, abnormal ECG, or a positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies
* If a woman, be pregnant, lactating or completed last term pregnancy within 6 months before admission to study center on Day -1
* Have known allergy to heparin (agent used to prevent clotting of the blood) or history of heparin induced thrombocytopenia (low blood platelet count as a result of the medication heparin)
* Have intermediate or low activity of CYP2D6 as determined by genetic testing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-08; Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters (area under the plasma concentration-time curve [AUC] and the maximum plasma concentration [Cmax]) of 31001074 with and without the coadministration of paroxetine | 0 to 72 hours after study drug administration on Day 1 and Day 13

SECONDARY OUTCOMES:
The number and type of adverse events and serious adverse events reported | From screening (up to 29 days before study drug administration) through 30 days after Day 16 (study completion) or at the time of early withdrawal from the study
Results from clinical laboratory tests performed | During screening (15 to 29 days before study drug administration) through Day 16 or at the time of early withdrawal from the study
Findings from electrocardiograms (ECGs) and vital signs measurements performed | During screening (15 to 29 days before study drug administration) through Day 16 or at the time of early withdrawal from the study
Findings from physical examinations performed | During screening (15 to 29 days before study drug administration) and on Day 16 or at the time of early withdrawal from the study
Columbia Suicide Severity Rating Scale (C-SSRS) scores to assess severity and track suicidal events during treatment | During screening (15 to 29 days before study drug administration) through Day 16 or at the time of early withdrawal from the study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Overland Park, Kansas, United States